CLINICAL TRIAL: NCT00644761
Title: A Multi-Center Phase 2, Open-Label Study to Evaluate the Pharmacokinetics of Tacrolimus and Cyclosporine When Co-Administered With Adefovir Dipivoxil 10 mg to Patients Post-Liver Transplantation
Brief Title: PK Study of Tacrolimus and Cyclosporine When Co-Administered With Adefovir Dipivoxil in Post-Liver Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Elsa Mondou, MD, Gilead Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-02-531
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Post-Liver Transplantation; Adefovir Dipivoxil; Tacrolimus; Cyclosporine
MeSH Terms: conditions — Hepatitis B | interventions — adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm 1 (Other): Adefovir dipivoxil 10 mg once daily with tacrolimus or cyclosporine for 14 days
  Interventions: Drug: Adefovir Dipivoxil

INTERVENTIONS:
Drug: Adefovir Dipivoxil — Adefovir dipivoxil 10 mg once daily for 14 days co-administered with tacrolimus or cyclosporine

SUMMARY:
Open-label pharmacokinetic drug interaction study.

DETAILED DESCRIPTION:
Multi-center, phase 2, open-label, sequential-cohort, drug interaction study. Cohort 1 subjects (tacrolimus and adefovir dipivoxil) were enrolled first. Based on the findings in Cohort 1, a decision was made on whether to enroll subjects in Cohort 2 (cyclosporine and adefovir dipivoxil)(i.e., if no interaction was observed in Cohort 1, Cohort 2 subjects would not be enrolled). Since no pharmacokinetic interaction was observed in Cohort 1, Cohort 2 was not enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Greater than or equal to 6 months post-liver transplantation
* Must be on a documented stable total daily dose of tacrolimus or cyclosporine for three months.
* Must have calculated creatinine clearance greater than or equal 50 mL/min (Cockcroft-Gault method).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-02; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
To evaluate pharmacokinetics of tacrolimus or cyclosporine when co-administered with adefovir dipivoxil 10 mg once daily to patients post-liver transplantation | 21 days

SECONDARY OUTCOMES:
To evaluate PK of ADV 10 mg once daily when co-administered with tacrolimus or cyclosporine in patients post-liver transplantation. To evaluate the safety of ADV 10 mg once daily, when co-administered with tacrolimus or cyclosporine for 14 days. | 21 days

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NYU Medical Center, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Mayo Clinic, Rochester, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor Research Institute, Dallas, Texas

REFERENCES:
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-02-531_synopsis.pdf